CLINICAL TRIAL: NCT00580489
Title: Efficacy and Adverse Events of Morphine and Fentanyl in an Aeromedical Setting
Brief Title: Lifeflight: Fentanyl Versus Morphine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Charles Emerman, MD, Professor of Emergency Medicine, Case Western Reserve SOM, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB06-00065
Record Dates: First submitted 2007-12-21; First posted 2007-12-24 (Estimated); Results first posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-07

CONDITIONS: Pain Relief; Adverse Events
Keywords: helicopter; aeromedical; pain relief; analgesia; fentanyl; morphine; adverse events
MeSH Terms: conditions — Agnosia | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm C Morphine (Active Comparator): Morphine given to trauma patients transported by helicopter
  Interventions: Drug: either fentanyl or morphine
- Arm D Fentanyl (Active Comparator): Fentanyl given to trauma patients transported by helicopter
  Interventions: Drug: either fentanyl or morphine

INTERVENTIONS:
Drug: either fentanyl or morphine — either morphine 4mg IV or fentanyl 50mcg IV

SUMMARY:
The study is exempt from informed consent by the MetroHealth Medical Center institutional review board (IRB), because two standards of care are used and there is no increased clinical risk to the patient due to the study. The researchers randomize either fentanyl or morphine to be given to trauma patients and record how their pain scale is treated along with observing for adverse events. They are looking to see if the hypothesized benefits of fentanyl (which is much more expensive than morphine) actually exist.

DETAILED DESCRIPTION:
Periodic reports are made to the IRB.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patient
* Able to speak/communicate a pain scale

Exclusion Criteria:

* Age <18
* Age >69
* Initially or any time hypotensive
* Prisoner

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Smith, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Smith MD, Wang Y, Cudnik M, Smith DA, Pakiela J, Emerman CL. The effectiveness and adverse events of morphine versus fentanyl on a physician-staffed helicopter. J Emerg Med. 2012 Jul;43(1):69-75. doi: 10.1016/j.jemermed.2011.05.018. PMID 21689900

RESULTS

PARTICIPANT FLOW:
Groups:
- Morphine: Patients randomized on even days received Morphine 4mg IV
- Fentanyl: Patients randomized on odd days received Fentanyl 50mcg IV
Period: Overall Study
Arm/Group | Morphine | Fentanyl
Started | 104 | 100
Completed | 104 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Morphine: morphine for trauma patients transported by helicopter
  either fentanyl or morphine: either morphine 4mg IV or fentanyl 50mcg IV
- Fentanyl: fentanyl for trauma patients transported by helicopter
  either fentanyl or morphine: either morphine 4mg IV or fentanyl 50mcg IV
- Total: Total of all reporting groups
Arm/Group | Morphine | Fentanyl | Total
Number analyzed (Participants) | 103 | 97 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (13) | 39 (13) | 38.5 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 77 | 74 | 151
Initial Numeric Pain Score [Mean (Standard Deviation); unit: units on a scale] — Numeric Pain Score (NPS) 0-10, 0 Least pain, 10 most pain
  units on a scale | 8.0 (2.0) | 8.0 (1.8) | 8.0 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Numeric Pain Score (NPS) From First to Last Dose
Description: Mean difference in the numeric pain score (NPS) from the first dose to the final dose of medication administered.
  A significant mean pain score change is defined as greater than or equal to 2
  Numeric Pain Score (NPS) 0-10, 0 Least pain, 10 most pain
Time Frame: Medication was administered over a mean transport time of 37 minutes in the Morphine group and 43 minutes in the Fentanyl group.
Population: 4 subjects were excluded from analysis, 1 from the Morphine Group and 3 from the Fentanyl group to achieve the baseline participants for data analysis 103 morphine and 97 fentanyl.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Morphine | Fentanyl
Number analyzed (Participants) | 103 | 97
score on a scale | 2.2 (2) | 2.5 (2.7)

2. Secondary Outcome: Recording of Instance of Narcotic Side Effects.
Description: Instances of narcotic side effects (vital sign derangement, itching, nausea/vomiting) .
Time Frame: Groups were observed a mean of 37 minutes in the Morphine Group and a mean of 43 minutes in the Fentanyl group for side effects.
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Arm C Morphine: Morphine given to trauma patients transported by helicopter
  morphine 4mg IV
- Arm D Fentanyl: Fentanyl given to trauma patients transported by helicopter
  fentanyl 50mcg IV
Arm/Group | Arm C Morphine | Arm D Fentanyl
Number analyzed (Participants) | 103 | 97
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 hour
Description: 4 subjects were excluded from analysis, 1 from the Morphine Group and 3 from the Fentanyl group to achieve the baseline participants for data analysis 103 morphine and 97 fentanyl.
Groups:
- Morphine 4 mg iv; Fentanyl 50mcg IV: either fentanyl or morphine
  either fentanyl or morphine: either morphine 4mg IV or fentanyl 50mcg IV
Arm/Group | Morphine 4 mg iv | Fentanyl 50mcg IV
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/97
Other Adverse Events (participants affected / at risk) | 0/103 | 0/97

LIMITATIONS AND CAVEATS:
Power of study may be too low to determine small differences

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes